CLINICAL TRIAL: NCT04804982
Title: Study of the Use of Hearing Protection Equipment in the Occurence of Acute Acoustic Trauma in the Army
Acronym: QPROTEC
Status: Completed | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PBMD06; 2020-A03519-30 (Other: IDRCB)
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Acoustic Trauma
MeSH Terms: conditions — Hearing Loss, Noise-Induced | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — The participants will have to fill in a questionnaire about their knowledge and their attitude regarding auditory risk.

SUMMARY:
Each year, military epidemiological surveillance counts approximately 1,000 acute acoustic injuries. Most are caused by exposure to weapon noise during training sessions while military personnel are provided with hearing protection. Several hypotheses could explain the occurrence of acute acoustic trauma despite wearing protections:

* A lack of practices or knowledge about the use of hearing protection equipment that could facilitate the occurrence of acute acoustic trauma (improper fitting, use of an inappropriate type of protection, dropping of protectors, inappropriate removal)
* A failure to seal the external ear canal due to an inappropriate plug size. These hypotheses will be explored using a questionnaire distributed to a population of Army soldiers training to shoot.

The main objective is to determine the predictive factors corresponding to practices or knowledge related to the use of hearing protection equipment in the occurrence of acute acoustic trauma in a population of Army soldiers.

ELIGIBILITY:
Inclusion Criteria:

* Be a member of the Army
* Having performed at least one shooting session in the last 12 months

Exclusion Criteria:

* Inability to read and/or write in French language

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will be composed of male and female Army soldiers practicing shooting on a regular basis.
Sampling Method: Non-Probability Sample
Enrollment: 394 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Measurement of the importance of variables corresponding to practices or knowledge related to the use of hearing protection equipment in the occurrence of acute acoustic trauma. | At enrollment
  The importance of variables will be measured thanks to a random forest algorithm.

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - 119e Antenne Médicale, 14e Centre Médical des Armées, Angers
  - 101e Antenne Médicale, 13e Centre Médical des Armées, Angoulême
  - Institut de Recherche Biomédicale des Armées, Brétigny-sur-Orge
  - 93e Antenne Médicale, 8e Centre Médical des Armées, Brive-la-Gaillarde
  - 176e Antenne Médicale, 11e Centre Médical des Armées, Montauban
  - 31e Antenne Médicale, Suippes
  - 76e Antenne Médicale, 7e Centre Médical des Armées, Varces-Allières-et-Risset

IPD SHARING:
Plan to Share IPD: Undecided